CLINICAL TRIAL: NCT03262376
Title: Acute Effect of Minerals and Botanicals in Combination or Isolation on Cognitive Performance, Neural Activity, and Subjective and Cortisol Response to Acute Stress
Brief Title: Minerals and Botanicals for Acute Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Prof Louise Dye, Professor of Nutrition and Behaviour, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IIT15073
Record Dates: First submitted 2017-08-14; First posted 2017-08-25 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Stress; Anxiety
Keywords: Stress; Anxiety; Cortisol; Vitamins; Botanicals; Minerals
MeSH Terms: conditions — Anxiety Disorders | interventions — Minerals; Vitamins

STUDY DESIGN:
Intervention Model Description: The study conforms to a double blind, quasi-randomised (randomisation will be balanced across condition based on age and sex), placebo controlled, parallel group design comprising 4 treatment conditions
Who Masked: Participant, Care Provider, Investigator
Masking Description: This study is double-blinded. The supplement manufacturer will independently create codes for the 4 treatment conditions. The study statistician will use the treatment codes generated to allocate participants to treatments. Researchers and participants will be blind treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mineral + vits + botanical A (Experimental): Mineral and vitamin complex combined with Botanical A
  Interventions: Dietary Supplement: Minerals + Vitamins; Dietary Supplement: Botanical A
- Mineral + vits + botanical B (Experimental): Mineral and vitamin complex combined with Botanical B
  Interventions: Dietary Supplement: Minerals + Vitamins; Dietary Supplement: Botanical B
- Mineral+vits +botanical A+Botanical B (Experimental): Mineral and vitamin complex combined with Botanical A and Botanical B
  Interventions: Dietary Supplement: Minerals + Vitamins; Dietary Supplement: Botanical A; Dietary Supplement: Botanical B
- Placebo (Placebo Comparator): Cellulose crystalline placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Minerals + Vitamins — A mineral and vitamin tablet
  Arms: Mineral + vits + botanical A; Mineral + vits + botanical B; Mineral+vits +botanical A+Botanical B
Dietary Supplement: Botanical A — Botanical extract administered in capsule form
  Arms: Mineral + vits + botanical A; Mineral+vits +botanical A+Botanical B
Dietary Supplement: Botanical B — Botanical extract administered in capsule form
  Arms: Mineral + vits + botanical B; Mineral+vits +botanical A+Botanical B
Other: Placebo — Cellulose crystalline tablet
  Arms: Placebo

SUMMARY:
The objective of this acute intervention study is to examine the potential of minerals combined with botanicals to demonstrate unique and synergistic effects on oscillatory brain activity, cognitive performance, and stress reduction (endocrine, sympathetic, and subjective parameters) under conditions of acute stress in moderately stressed individuals

DETAILED DESCRIPTION:
Botanicals in isolation or combined, will be administered with a mineral and vitamin complex to moderately stressed, healthy adults in a parallel groups fashion in this randomised placebo controlled trial. Oscillatory brain activity (EEG) during rest and performance on cognitive tasks of attention will be examined after treatment intake under conditions of acute laboratory stress. The effects of treatments on stress responses (cardiovascular, subjective and cortisol responses) will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Adults capable of giving informed consent
* Male and Female
* ≥18 - ≤50 years of age (premenopausal if female)
* Effective contraception taken in females
* Women in luteal menstrual phase
* Body mass index (BMI) ≥18 and ≤30 kg/m2
* Normal vision or corrected to normal
* Moderately stressed (subjective report)

Exclusion Criteria:

* No known intolerance to minerals, vitamins or botanicals
* Intake of prescribed medication except contraceptives
* Intake of any regular medication/supplements
* History of significant hypertensive, hepatic, renal, pulmonary, gastro-intestinal, endocrinological, neurologic, haematological, psychiatric (inc. mood disorders), cardiac or allergic disease which is clinically relevant to the study
* Hypertension (self-report or resting blood pressure >160/95 mmHg)
* Diabetes (T1 or T2)
* Smoking more than occasional cigarettes (>5/day)
* Pregnant or lactating
* Previous participation in a stress study involving the Trier Social Stress Test
* Night-working/shift work
* Recreational drug use

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
Oscillatory brain activity during the rested state and attentional processing (EEG; Biosemi Active2, 64-channel, DC amplifier, 24-bit resolution system) | 30 minute period, approximately 65 minutes post treatment intake
  The effect of treatment on oscillatory brain activity during the rested state and during attentional task processing after stress exposure

SECONDARY OUTCOMES:
Subjective stress (Stress & Arousal Checklist; Mackay et al., 1978) | Acute responses to stress induction from pre-treatment intake to approximately 8 hours post-treatment intake
  The effect of treatment on subjective stress responses to stress induction
Subjective mood (Profile of Mood States [MCNair et al., 1971] & Bond Visual analogue scales, 1974) | Acute responses to stress induction from pre-treatment intake to approximately 8 hours post-treatment intake
  The effect of treatment on subjective mood responses to stress induction
Subjective anxiety (Spielberger State Trait Anxiety Inventory, 1983) | Acute responses to stress induction from pre-treatment intake to approximately 8 hours post-treatment intake
  The effect of treatment on subjective anxiety responses to stress induction
Cognitive performance (Digit attention switching & threat vs neutral dot probe task) | 20 minute period (comprising two distinct tasks) approximately 75 minutes post treatment intake
  The effect of treatment on reaction time and accuracy performance on two cognitive tasks of attention
Blood pressure | Acute responses to stress induction from pre-treatment intake to approximately 8 hours post-treatment intake
  The effect of treatment on blood pressure responses to stress induction
Heart rate | Acute responses to stress induction from pre-treatment intake to approximately 8 hours post-treatment intake
  The effect of treatment on heart rate variability before and after stress induction
Salivary cortisol | Acute responses to stress induction from pre-treatment intake to approximately 8 hours post-treatment intake
  The effect of treatment on salivary cortisol responses to stress induction
Event related potentials (EEG; Biosemi Active2, 64-channel, DC amplifier, 24-bit resolution system) | 20 minute period (comprising two distinct tasks) approximately 75 minutes post treatment intake
  The effect of treatment on event related potentials during execution of attentional processing

CONTACTS AND LOCATIONS:
Overall Officials: Louise Dye, PhD, Principal Investigator — University of Leeds
Locations (1):
- Human Appetite Research Unit, University of Leeds, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boyle NB, Dye L, Lawton CL, Billington J. A Combination of Green Tea, Rhodiola, Magnesium, and B Vitamins Increases Electroencephalogram Theta Activity During Attentional Task Performance Under Conditions of Induced Social Stress. Front Nutr. 2022 Jul 22;9:935001. doi: 10.3389/fnut.2022.935001. eCollection 2022. PMID 35938130
- [Derived] Boyle NB, Billington J, Lawton C, Quadt F, Dye L. A combination of green tea, rhodiola, magnesium and B vitamins modulates brain activity and protects against the effects of induced social stress in healthy volunteers. Nutr Neurosci. 2022 Sep;25(9):1845-1859. doi: 10.1080/1028415X.2021.1909204. Epub 2021 Apr 26. PMID 33896388